CLINICAL TRIAL: NCT05755984
Title: 3D Printed Breast Models in the Surgical Management of Breast Cancer
Status: Suspended | Phase: Not Applicable | Type: Interventional
Why Stopped: DMC Monitor Action
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: University Cancer Foundation via the Institutional Research Grant program at the University of Texas MD Anderson Cancer Center (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2021-1201; NCI-2023-01852 (Other: NCI-CTRP Clinical Trials Registry)
Record Dates: First submitted 2023-02-20; First posted 2023-03-06 (Actual); Last update posted 2026-02-02 (Actual); Status verified 2026-01

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arm 1: 3D printed model (Experimental): a 3-D printed model of your breast will be created and discussed with participants during your surgical consultation.
  Interventions: Diagnostic Test: 3D printed model
- Arm 2: No 3D printed model (No Intervention): Participants will have a standard-of-care surgical consultation using traditional breast imaging.

INTERVENTIONS:
Diagnostic Test: 3D printed model — scan
  Arms: Arm 1: 3D printed model

SUMMARY:
To learn if providing a 3-D printed model of the breast can help breast cancer patients make decisions related to their care. During this study, some study participants will receive the 3-D printed model and some study participants will receive traditional breast imaging scans to learn if the 3-D printed model

DETAILED DESCRIPTION:
Primary Objective:

•The objective of this prospective study is to determine the impact of 3D printed breast models, compared to 2D imaging, on breast cancer patients' decisional conflict related to treatment decision-making.

Secondary Objective:

* To observe if patients will change their initial desired surgical option (mastectomy versus lumpectomy) after viewing the 3D printed models
* To evaluate the quality of the communication between surgical providers and patients with and without the 3D printed models
* To assess the surgical outcome including the margin status
* To evaluate patient satisfaction and well-being post-surgery between the 3D printed model group and the control group as well as mastectomy versus lumpectomy subgroups
* To assess surgical providers' response to the acceptability and utility of the model

ELIGIBILITY:
Inclusion Criteria:

* Age 18 or older female
* Patient must have histologically confirmed breast malignancy
* Patient is a candidate for surgical management
* Patient has a surgeon at MDACC (main campus and/or Houston Area Locations)
* Patient has a breast MRI for extent of disease assessment at MDACC (main campus and/or Houston Area Locations).
* Patient is able to speak, read or write English
* Patient is willing to be randomized to the control or 3D printed breast model groups and is willing to sign the consent form.

Exclusion Criteria:

* Pregnant and breastfeeding patients
* Patients who had history of mastectomy, have recurrent malignancies on the mastectomy side
* Patients for whom it is not feasible to create a 3D printed breast model from breast MRI

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2024-02-29 (Actual); Primary Completion 2026-02-28 (Estimated); Study Completion 2028-02-28 (Estimated)

PRIMARY OUTCOMES:
Decision Conflict Scale (DCS) score questionnaires | through study completion; an average of 1 year.
  Score scale ranges: Strongly Agree 1, Agree 2 Neither agree or Agree 3 Strongly Disagree 4

CONTACTS AND LOCATIONS:
Overall Officials: Lauren Chang Sen, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- M D Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: M D Anderson Cancer Center — http://www.mdanderson.org